CLINICAL TRIAL: NCT02326467
Title: Pilot Study: Safety of Chlorhexidine (CHG) Baths in Patients Less Than 2 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celeste Chandonnet (Other)
Responsible Party: Sponsor-Investigator, Celeste Chandonnet, Unit based Infection Prevention Nurse, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00011128
Record Dates: First submitted 2014-06-25; First posted 2014-12-29 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Chlorhexidine Allergy; Infection; Rash
Keywords: chlorhexidine; safety; bath; rash; infant
MeSH Terms: conditions — Infections; Exanthema | interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chlorhexidine gluconate bath (Experimental): All subjects will receive a bath twice a week with 2% CHG bathing cloths. The baths will be followed by blood sampling for CHG levels prior to initiation of baths and every Friday for the duration of study participation. The study team will monitor the infant's skin for evidence of untoward lesions prior to the first bath and every 12 hours during the course of the study. CHG blood levels will be monitored for associated adverse events and accumulation.
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Bi-weekly chlorhexidine baths
  Other Names: Sage® 2% Chlorhexidine Gluconate Cloth

SUMMARY:
Literature provides overwhelming evidence supporting the use of chlorhexidine gluconate (CHG) a rapid onset, broad spectrum, topical antiseptic for reducing healthcare-associated infections (HAIs). CHG is believed to be superior to other forms of antiseptics because, when it is applied to the skin surface, it leaves a lasting residue on the skin. CHG has been shown to be well tolerated in patients 2 months of age and older. However there is limited evidence to support the use of topically applied CHG in infants less than 2 months of age because of potential safety concerns in this population. The purpose of this study will be to describe the safety of bi-weekly CHG baths in a sample of Newborn Intensive Care Unit (NICU) and pediatric Cardiac Intensive Care Unit (CICU) patients by measuring the incidence of skin problems and CHG blood levels.

DETAILED DESCRIPTION:
Evidence overwhelmingly supports the use of Chlorhexidine Gluconate (CHG) a rapid onset, broad spectrum, topical antiseptic for reducing Healthcare-associated Infections (HAIs). CHG provides prolonged protection against both gram-positive and gram-negative organisms. Reports indicate CHG is well tolerated in patients greater than two months of age. However, due to safety concerns, there is limited evidence to support the use of topically applied CHG in infants less than 2 months of age.

The purpose of this Phase I Clinical (pilot) study is to describe the safety of bi-weekly CHG baths in a sample of 50 Newborn Intensive Care Unit (NICU) and pediatric Cardiac Intensive Care Unit (CICU) patients, (36 weeks PMA or older, less than 2 months of age or 48 weeks PMA and with a CVC), by measuring the incidence of skin problems and CHG blood levels. CHG baths will be performed every Monday and Thursday during the day shift, for up to 12 weeks post enrollment or until the CVC is removed or the patient is discharged.

Chlorhexidine Gluconate bathing cloths are marketed for peri-operative skin preparation. However, daily CHG baths are a common practice in ICUs around the nation because of its proven method for preventing HAIs in patients > 2 months of age and older. Furthermore, CHG use for skin antisepsis has become a widely accepted practice, and it is now part of the Centers for Disease Control and Prevention (CDC) CVC maintenance bundle for use in patients greater than 2 months of age, and a recommendation to use with caution in infants < 2 months of age.

Hypothesis 1:CHG will be safe for use in a sample of infants 36 weeks PMA or older, and less than 2 months of age (48 weeks PMA) with a CVC as evidenced by an adverse event rate less than 10%.

Hypothesis 2: Twice weekly CHG baths do not lead to rising (cumulative) CHG blood levels, LFTs (AST/ALT) and Serum Creatinine over time in a sample of infants 36 weeks PMA or older, and less than 2 months of age (48 weeks PMA) with a CVC..

ELIGIBILITY:
Inclusion criteria.

* Greater than/equal to 36 weeks PMA (gestational age + chronological age)
* Less than/equal to 48 weeks PMA (gestational age + chronological age)
* Greater than/equal to 3 days of age
* Existing or soon to be placed, peripheral or surgical CVC
* Permission to participate in trial by attending physician
* Parent or legal guardian informed consent to participate in the trial

Exclusion criteria.

* • Infant with a large open lesion or severe skin condition (i.e., Myelomeningocele, Gastroschisis, lymphatic malformation, open chest, ostomies and/or mucus fistulas or Icthyosis)
* Infants with active seizure disorders
* Infants with Hypoxic Ischemic Encephalopathy
* Infants with severe multi-system organ failure or Liver failure as defined by documentation of abnormal liver function tests: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) Gamma-glutamyltransferase (GGT) and L-lactate dehydrogenase (LD).
* Infant with renal impairment as defined by: documented serum Creatinine greater than 0.7, renal disorders (renal agenesis, polycystic kidney disease, dysplastic kidneys, acute renal injury).
* Infants deemed clinically unstable by their physician such as patients that are extremely fragile and wouldn't tolerate the stimulation of the bathing process or those infants being considered for withdrawal of care.

Ages: 36 Weeks to 48 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste J Chandonnet, BSN CCRN CIC, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the ten subjects enrolled, one subject withdrew prior to any interventions per parental request.
Groups:
- Chlorhexidine Gluconate Bath: All subjects were to receive a bath twice a week with 2% CHG bathing cloths. The baths were to be followed by blood sampling for CHG levels prior to initiation of baths and every Friday for the duration of study participation. The study team monitored the infant's skin for evidence of untoward lesions prior to the first bath and every 12 hours during the course of the study. CHG blood levels were to be monitored for associated adverse events and accumulation.
  Chlorhexidine gluconate: Bi-weekly chlorhexidine baths
Period: Overall Study
Arm/Group | Chlorhexidine Gluconate Bath
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Chlorhexidine Gluconate Bath: All subjects received a bath twice a week with 2% CHG bathing cloths. The baths were to be followed by blood sampling for CHG levels prior to initiation of baths and every Friday for the duration of study participation. The study team monitored the infant's skin for evidence of untoward lesions prior to the first bath and every 12 hours during the course of the study. CHG blood levels were to be monitored for associated adverse events and accumulation.
  Chlorhexidine gluconate: Bi-weekly chlorhexidine baths
Arm/Group | Chlorhexidine Gluconate Bath
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: Weeks]
  PMA (Weeks) | 40 [36 to 43.7]
Age, Continuous [Median (Full Range); unit: Age (Days)] | 21 [4 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Weight Demographics [Median (Full Range); unit: Grams]
  Birth Weight | 2840 [1625 to 3880]
  Weight at Enrollment | 2840 [1670 to 3880]
Type of Central Venous Line [Count of Participants; unit: Participants]
  PICC | 6
  Broviac | 1
  Umbilical | 1
  Right Atrium | 1
Diagnosis [Count of Participants; unit: Participants]
  Coarctation of the Aorta | 1
  Duodenal Atresia | 1
  Esophageal Atresia | 1
  Esophageal Atresia/Tracheal Esophageal Fistula | 1
  Gastroschisis | 2
  Hypoplastic Left Heart Syndrome | 1
  Laryngeal Cleft (Type III) | 1
  Transposition of the Great Arteries | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Study Participants With Skin Reactions Less Than 10%
Description: 1. Study RN's will perform a full body skin assessment for skin irritation or open areas prior to each bath.
  2. Bedside RN's will complete skin assessments every 12 hours during the course of the study.
  3. Descriptive statistics including mean, median, range and frequencies will be used to describe adverse events (including skin reactions and other untoward events). We will characterize the demographic and clinical characteristics of subjects that experience adverse events, although we will not perform hypothesis tests of association. We will consider time-to-rash data using Kaplan-Meier estimators.
Time Frame: Adverse Events assessed every 12 hours for the duration of study participation (max 90 days)
Population: All subjects were observed for adverse skin reactions related to CHG bathing.
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Bath
Number analyzed (Participants) | 9
Participants
  AE Skin Reactions | 0
  AE Anemia | 2

2. Secondary Outcome: The Number of Participants With Detectable CHG Blood Levels
Description: To monitor for absorption into the blood, a single CHG level will be obtained at baseline and then weekly on Fridays for the remainder of the study for each study participant. A CHG level will also be drawn when an infant is removed from the study in response to an adverse reaction. Of note, a threshold for safe, normal or toxic CHG level is not known, thus we will closely monitor blood levels and convene a meeting of the Data Safety and Monitoring Committee (DSMC) if adverse reactions develop in association with elevated blood levels.
Time Frame: CHG blood levels will be assessed at baseline, then weekly for the duration of study participation (max 90 days)
Population: CHG levels were recorded in all participants.
Measure: Count of Participants; unit: Participants
Groups:
- Chlorhexidine Gluconate Bath: All subjects received a bath twice a week with 2% CHG bathing cloths. The baths were followed by blood sampling for CHG levels prior to initiation of baths and every Friday for the duration of study participation. The study team monitored the infant's skin for evidence of untoward lesions prior to the first bath and every 12 hours during the course of the study. CHG blood levels were monitored for associated adverse events and accumulation.
  Chlorhexidine gluconate: Bi-weekly chlorhexidine baths
Arm/Group | Chlorhexidine Gluconate Bath
Number analyzed (Participants) | 9
Participants
  Participants with non-detectable CHG levels or CHG levels < 100 ng/mL for duration of study. | 2
  Participants with highest recorded CHG level equal to or < 1000 ng/mL for duration of study. | 4
  Participants with highest recorded CHG level > 1000 ng/mL for duration of study. | 3

ADVERSE EVENTS:
Time Frame: The adverse event data collection period for enrolled subjects were collected up to a maximum of 40 days.
Description: All subjects were monitored for adverse events including skin reactions, anemia and significant changes to baseline lab values.
Arm/Group | Chlorhexidine Gluconate Bath
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorhexidine Gluconate Bath (N=9)
Anemia (Blood and lymphatic system disorders) | 2 (2) — One subject experienced anemia that was identified with pre-operative lab work. The subject was placed on study hold for anemia and post-op recovery. The anemia resolved post-op. This was not deemed a serious adverse event.

LIMITATIONS AND CAVEATS:
The study was stopped early due to the unknown risks associated with CHG levels in relation to CHG bathing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02326467/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT02326467/ICF_001.pdf